CLINICAL TRIAL: NCT05806502
Title: The Effect of Arginase Inhibition on Vascular Endothelial Function in Patients With Type 1 and Type 2 Diabetes
Brief Title: Arginase Inhibition in Type 1 and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, Principal investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T1DM study
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 diabetes (Experimental): Endothelium-dependent and -independent vasodilatation before and after 120 min intra-arterial administration of arginase the inhibitor N-omega-hydroxy-nor-l-arginine (nor-NOHA).
  Interventions: Diagnostic Test: Nω-hydroxy-nor-arginine
- Type 2 diabetes (Experimental): Endothelium-dependent and -independent vasodilatation before and after 120 min intra-arterial administration of arginase the inhibitor N-omega-hydroxy-nor-l-arginine (nor-NOHA).
  Interventions: Diagnostic Test: Nω-hydroxy-nor-arginine

INTERVENTIONS:
Diagnostic Test: Nω-hydroxy-nor-arginine — Arginase inhibitor

SUMMARY:
To evaluate the efficacy of arginase inhibition on endothelial function in patients with type 1 diabetes and type 2 diabetes.

DETAILED DESCRIPTION:
Detailed Description:

The study is performed on one group of patients with type 1 diabetes and one group of patients with type 2 diabetes.

Forearm blood flow is determined by venous occlusion plethysmography. Endothelium-dependent vasodilatation is determined during intra-brachial artery infusion of serotonin (21, 70 and 210 ng/min). Endothelium-independent vasodilatation is determined by infusion of sodium nitroprusside (SNP; 1, 3 and 10 µg/min). Each dose is given for 2 min at a rate of 2.5 ml/min. Data are expressed as percentage change in forearm blood from baseline flow.

Twelve subjects are included in each group. On the day of the study the subject arrives to the laboratory after having a light breakfast. Forearm vessels of the non-dominant arm are cannulated and forearm blood flow is determined as described above. Baseline endothelium-dependent and endothelium-independent vasodilatation is determined by intra-arterial infusions of serotonin and SNP, respectively. Thereafter an intra-arterial infusion of the arginase inhibitor N-omega-hydroxy-nor-l-arginine (nor-NOHA) is administered as an intra-arterial infusion at a rate of 0.1 mg/min and is maintained for 120 min. The dose is based on a previous study by our group demonstrating improved endothelial function. Endothelium-dependent and -independent vasodilatation is reassessed at 120 min of infusion.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes

Exclusion Criteria:

* Age >80 years
* Acute coronary or ischemic event during the last three months
* Vascular surgery of the arm
* Peripheral vascular disease affecting the arm
* Ongoing anticoagulant medication
* Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Endothelium-dependant increase in forearm blood flow | 120 minutes
  Change in forearm blood flow

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden